CLINICAL TRIAL: NCT02505243
Title: Evaluation of RIBAvirin Plasma COncentrations in Patients With Chronic Hepatitis C Infection Routinely Treated With Modern DAA Regimens
Acronym: RIBACOP
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other); University Medical Center Groningen (Other); UMC Utrecht (Other); Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCN-AKF-15.03
Record Dates: First submitted 2015-07-15; First posted 2015-07-22 (Estimated); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: HCV Coinfection; Hepatitis C
Keywords: ribavirin; direct-acting antivirals; pharmacokinetics; therapeutic drug monitoring
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HCV patients: HCV patients treated with direct acting antivirals and ribavirin

SUMMARY:
The aim of this study is to evaluate RBV plasma concentrations when used in combination with newly developed DAA combinations. If possible, its correlations with SVR rates and incidence of anaemia will be assessed in HCV-patients.

DETAILED DESCRIPTION:
Ribavirin (RBV) is a synthetic guanosine analogue that is used to treat patients infected with hepatitis C virus (HCV). For many years, RBV has been the cornerstone of the HCV treatment in combination with peg interferon (PEG-IFN). Since the development of direct-acting antivirals (DAA), PEG-IFN free treatment regimes became first choice of HCV treatment in the Netherlands. RBV still plays an important role in some of these regimens. The European Association for the Study of the liver (EASL) included RBV in PEG-IFN free regimens in combination with sofosbuvir, simeprevir and daclatasvir for HCV genotype (GT) 1, 3 and 4. Patients with predictors of poor response are candidates for DAA therapy combined with RBV, for instance prior null responders and/or patients with cirrhosis. For the treatment of genotype 2 (GT2) and 3 RBV is used in combination with sofosbuvir.

Chronic HCV infection is treated with combination therapy, therefore manufacturers developed combination tablets such as Gilead's Harvoni (ledipasvir + sofosbuvir) and Abbvie's 3D combination (paritaprevir, ombitasvir, dasabuvir and ritonavir). Possibly, RBV will be added to these regimes in the future when the patient is a prior null responder or suffering from cirrhosis.

As RBV is a guanine analogue it is not specific for HCV and some severe adverse effects are known. The most important adverse effect is haemolytic anaemia,which usually occurs during the first weeks of treatment (>10% of the treated patients, depending on co-medication). Other adverse reactions that were frequently reported were: neutropenia, anorexia, depression/insomnia, headache, dizziness, dyspnea, and cough 5.

In dual (PEG-IFN + RBV) HCV therapy RBV concentrations were associated with efficacy and toxicity. Also in former studies in HCV-infected patients treated with telaprevir (TVR) or boceprevir (BOC) in combination with PEG-IFN, the plasma concentration of RBV was associated with Sustained Virologic Response (SVR) and anaemia (defined as Hb<8,5 g/dL). We have tried to determine an optimal therapeutic range for RBV when combined with these DAAs. The plasma concentration of RBV at week 8 should be 2.2-5.3 mg/L in combination with TVR. 48% of the HCV patients in the cohort had these plasma concentrations of which 81% achieved SVR and 5.2% reported anaemia. In combination with BOC the plasma concentration should be 2.2-3.6 mg/L, 50% of patients had these concentrations. In this group 69% of patients achieved SVR and 46% anaemia. So, for these therapies, therapeutic ranges for RBV could be defined for the optimal SVR rates and the lowest incidence of anaemia 6, 7.

As TVR and BOC have now been replaced by novel DAAs, we would like to investigate this described relationship between RBV concentrations, SVR and anaemia also with the newer DAAs that were licensed in the last year (simeprevir and sofosbuvir) and that are going to be available in 2015 in The Netherlands (daclatasvir, Harvoni, Abbvie 3D combo).

The aim of this study is to evaluate RBV plasma concentrations when used in combination with newly developed DAA combinations. If possible, its correlations with SVR rates and incidence of anaemia will be assessed in HCV-patients.

ELIGIBILITY:
Inclusion Criteria:

* HCV-infected patients
* Patient must be treated with ribavirin. The dosage of ribavirin may vary, as the different centers have different protocols for RBV dosing.
* Patient must be treated with one or more DAAs (simeprevir, sofosbuvir, daclatasvir, ledipasvir, paritaprevir, ombitasvir, or dasabuvir).
* At least 18 years of age at start of treatment.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: chronicHCV infected patients treated with direct acting antivirals (daclatasvir, simeprevir, sofosbuvir, paritaprevir, ombitasvir, dasabuvir, ledipasvir) and ribavirin.
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2015-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Ribavirin concentration | Ribavirin concentraition at week 8 of treatment
  Analysis ribavirin concentration in plasma

SECONDARY OUTCOMES:
Sustained virological response (SVR12) | Change from baseline virological resonse, 12 weeks after treatment.
  HCV RNA analysis in plasma
Hemoglobin concentrations | Change from baseline hemoglobin concentrationes, 8 weeks after treatment.
  Analysis Hb plasma concentration
Ribavirin concentration | Ribavirin concentraition at week 2 of treatment
  Analysis ribavirin concentrations in plasma

CONTACTS AND LOCATIONS:
Overall Officials: David Burder, PharmdD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Result] van Tilborg M, Lieveld FI, Smolders EJ, van Erpecum KJ, de Kanter CTMM, Maan R, van der Valk M, Arends JE, Dofferhoff ASM, Blokzijl H, Bijmolen M, Drenth JPH, de Knegt RJ, Burger DM; HepNed Study Group. Ribavirin steady-state plasma level is a predictor of sustained virological response in hepatitis C-infected patients treated with direct-acting antivirals. Aliment Pharmacol Ther. 2017 Nov;46(9):864-872. doi: 10.1111/apt.14288. Epub 2017 Sep 7. PMID 28881031